CLINICAL TRIAL: NCT07400263
Title: A Prospective Clinical Study of an EpCAM-Targeted Radiotracer for Molecular Imaging of Epithelial Tumors
Brief Title: Evaluation of an EpCAM-Targeted Radiotracer in Epithelial Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xing Yang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025PHB625
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Epithelial Tumors, Malignant
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EpCAM PET (Experimental)
  Interventions: Diagnostic Test: [68Ga]Ga-PN-EpC1 PET/CT

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-PN-EpC1 PET/CT — Participants will receive a single intravenous administration of the EpCAM-targeted radiotracer [68Ga]Ga-PN-EpC1 for PET/CT imaging. The radiotracer will be administered at a dose of 0.05-0.1 mCi/kg, followed by whole-body PET/CT acquisition according to the study imaging protocol. Additional dynamic or delayed imaging may be performed in selected participants.

SUMMARY:
The goal of this prospective, single-arm clinical trial is to evaluate the imaging performance and safety of an EpCAM-targeted radiotracer, [68Ga]Ga-PN-EpC1, in patients with epithelial tumors.

The main questions it aims to answer are:

* What is the sensitivity of [68Ga]Ga-PN-EpC1 PET/CT for detecting EpCAM-positive tumor lesions?
* How does the radiotracer uptake correlate with EpCAM expression assessed by immunohistochemistry?
* Is [68Ga]Ga-PN-EpC1 safe and well tolerated when administered for PET/CT imaging in patients with epithelial tumors? Participants will undergo [68Ga]Ga-PN-EpC1 PET/CT imaging prior to tumor biopsy or surgical resection. Imaging findings will be analyzed and compared with histopathological results and standard imaging assessments. Safety will be evaluated by monitoring adverse events following radiotracer administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed or suspected tumors visiting the hospital between January 2026 and December 2026, who are scheduled for pathological biopsy or surgical treatment within 2 months.
2. Age > 18 years, regardless of gender.
3. Adequate organ and bone marrow function as defined by the following laboratory values:

   * Hematology: WBC ≥4.0×10^9/L or ANC ≥1.5×10^9/L; PLT ≥100×10^9/L; Hemoglobin ≥90 g/L.
   * Liver Function: Total bilirubin ≤1.5× ULN; ALT and AST ≤2.5× ULN (or ≤5× ULN if liver metastases are present).
   * Renal Function: BUN ≤1.5× ULN; Serum Creatinine (SCr) ≤1.5× ULN.
4. Normal cardiac function.
5. Expected life expectancy ≥12 weeks.
6. Presence of at least one measurable target lesion according to RECIST v1.1 criteria.
7. Patients recommended by clinicians to undergo PET/CT examination for tumor diagnosis and staging.
8. Women of childbearing potential must have a negative pregnancy test within 7 days prior to the examination. Male and female patients of reproductive age must agree to use effective contraception during the study and for at least 3 months after the examination.
9. Voluntarily participate in the study, demonstrate full understanding of the protocol, and provide written informed consent.

Exclusion Criteria:

1. Severe laboratory abnormalities, including significant impairment of hepatic or renal function, or severe hematological dysfunction.
2. History of allergic diseases.
3. Patients planning for pregnancy during the study period.
4. Pregnant or lactating women.
5. Inability to maintain a supine position for at least 30 minutes.
6. Patients with claustrophobia or other diagnosed psychiatric disorders that may interfere with compliance.
7. Any other condition that, in the opinion of the investigator, may increase the risk to the subject or interfere with the evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of [68Ga]Ga-PN-EpC1 PET/CT for lesion detection | From PET/CT imaging to histopathological confirmation within 2 months.
  Sensitivity of [68Ga]Ga-PN-EpC1 PET/CT for detecting epithelial tumor lesions, using histopathological results as the reference standard.

SECONDARY OUTCOMES:
Specificity and Accuracy of [68Ga]Ga-PN-EpC1 PET/CT for Lesion Detection | From PET/CT imaging to histopathological confirmation within 2 months.
  The specificity and overall diagnostic accuracy of [68Ga]Ga-PN-EpC1 PET/CT in identifying epithelial tumor lesions, using histopathological results as the reference standard.
Correlation Between [68Ga]Ga-PN-EpC1 Uptake and EpCAM Expression Levels | From PET/CT imaging to IHC analysis of biopsy or surgical specimens (within 2 months).
  To evaluate the correlation between the intensity of tracer uptake (e.g., SUVmax, SUVmean) on PET/CT images and the expression level of EpCAM in tumor tissues as determined by immunohistochemistry (IHC).
Safety of [68Ga]Ga-PN-EpC1 PET/CT Imaging | Within 72 hours post-injection of [68Ga]Ga-PN-EpC1.
  Assessment of the incidence and severity of adverse events (AEs) related to the administration of [68Ga]Ga-PN-EpC1, monitored via vital signs and patient reporting.

OTHER OUTCOMES:
Comparative Diagnostic Performance: Standard Structural Imaging vs. [68Ga]Ga-PN-EpC1 PET/CT | From initial imaging assessment to the end of follow-up at 2 years.
  Comparison of diagnostic efficacy (sensitivity, specificity, accuracy) between conventional imaging (e.g., CT, MRI, FDG PET/CT) and [68Ga]Ga-PN-EpC1 PET/CT at the patient-level, region-level, and lesion-level.
Optimal Cut-off Value of [68Ga]Ga-PN-EpC1 Uptake for Predicting Tumor Lesions | From PET/CT imaging to the end of follow-up at 2 years.
  To determine the optimal threshold (cut-off value) of PET semi-quantitative parameters (e.g., SUV max) for distinguishing malignant from benign lesions using Receiver Operating Characteristic (ROC) curve analysis.
Correlation of Tracer Uptake and Total Tumor Burden with Patient Prognosis | From PET/CT imaging to the end of follow-up at 2 years.
  To explore the association between [68Ga]Ga-PN-EpC1 PET/CT parameters (uptake intensity, tumor volume) and patient outcomes, such as Progression-Free Survival (PFS) or Overall Survival (OS).